CLINICAL TRIAL: NCT07079007
Title: Use of Water Ingestion to Improve Visualisation in Small Intestine Ultrasound (WIVIUS): Single Centre Blinded Crossover Trial
Brief Title: Use of Water Ingestion in Small Intestine Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Sheng Wei Lo, Principal Investigator: Julien Schulberg, MBBS, PhD , Austin Health, Melbourne, Austin Health
Other Study IDs: HREC/25015/Austin-2025
Record Dates: First submitted 2025-06-30; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Crohn Disease (CD); Intestine Ultrasonography
Keywords: small bowel contrast ultrasound
MeSH Terms: conditions — Crohn Disease | interventions — Water

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IUS oral contrast: All patients already referred and scheduled to undertake an IUS in the single-centre IUS clinic would undergo a baseline procedure. Patients that meet the inclusion and exclusion criteria would be asked to ingest 1000ml water as part of standard of care.
  Inclusion Criteria
  All consecutive patients at baseline scan with:
  Confirmed or suspected Crohn's disease with small bowel involvement Increased bowel wall thickness (>3mm) of the terminal ileum Suboptimal luminal distension of the terminal ileum 3cm proximal to ICV and 1cm proximal to diseased segment (defined as <8mm) All patients with an ileo-colic anastomosis
  Exclusion Criteria
  Presence of an ostomy Adequate distension at baseline scan Patients with ileo-rectal anastomosis or IPAA
  Interventions: Other: Water

INTERVENTIONS:
Other: Water — Patients that meet the inclusion and exclusion criteria would be asked to ingest 1000ml water as part of standard of care.

SUMMARY:
Small Intestine Contrast Ultrasonography (SICUS) is an ultrasound-based method that explores bowel loops, and is able to identify wall thickness, intestinal motility, bowel wall vascularity and complications such as stenosis or dilatation. Previous studies have utilised oral ingestion of an oral contrast solution (usually PEG dissolved in a volume of water ranging from 250 to 1000mL), in order to increase the sensitivity of ultrasound, especially in stricture detection. Parameters that have been improved include lumen distension to better delineate bowel wall layers, and improved peristalsis. Diffusion of this technique has been limited, in part due to PEG-based agents being costly, time consuming and are not tolerated well in some individuals. Utilisation of water as oral contrast may improve patient tolerability and therefore increase uptake of water ingested intestinal contrast ultrasound (WICUS) as a technique in routine clinical practice. The investigators aim to study the tolerability and the improvement of image quality utilising water as an oral contrast for intestinal ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients at baseline scan with:

* Confirmed or suspected Crohn's disease with small bowel involvement
* Increased bowel wall thickness (>3mm) of the terminal ileum
* Suboptimal luminal distension of the terminal ileum 3cm proximal to ICV and 1cm proximal to diseased segment (defined as <8mm)
* All patients with an ileo-colic anastomosis

Exclusion Criteria:

* Presence of an ostomy
* Adequate distension at baseline scan
* Patients with ileo-rectal anastomosis or IPAA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients already referred and scheduled to undertake an IUS in the single-centre Austin Health IUS clinic would undergo a baseline procedure. Patients that meet the inclusion and exclusion criteria would be asked to ingest 1000ml water as part of standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Improvement of luminal distension of the terminal ileum | At the post-water ingestion scan 20-30 minutes after ingestion
  Improvement of luminal distension of the terminal ileum, defined as increase of 20% over baseline luminal diameter at the terminal ileum if no disease, taking the average as measured at 1cm intervals over 3cm of the TI in longitudinal view. If diseased segment is present, then measurements would be done at 1cm intervals over 3cm proximal to the diseased segments.

SECONDARY OUTCOMES:
Is image quality and visualisation of the terminal/distal ileum improved post water ingestion during intestinal ultrasound compared to baseline as assessed by blinded sonographers | At the time of post-water ingestion scan 20-30 minutes after ingestion
  Recordings of the IUS would be recorded and de-identified
  Pre-contrast Cineloop x 1 of 10second duration encompassing the caecum, ileocaecal valce, terminal ileum extending to distal ileum
  Post-contrast Cineloop x 1 of 10second duration encompassing the caecum, ileocaecal valce, terminal ileum extending to distal ileum
  De-identified cineloops will then be randomised in a paired fashion (2 x cineloops baseline and 2 x cineloops post-contrast), and 3 external blinded sonographers will then be invited to review the cineloops - no limitation to number of times - and complete a questionnaire.
  Based on before and after CINE look in random order Global (overall image) assessment. Options: Better / Unchaged / Worse of CINEloop 1 compared to CINEloop 2

OTHER OUTCOMES:
Grade of peristalsis | At the time of post-water ingestion scan 20-30 mins after ingestion
  At the time of scan, determine grade of peristalsis (hyperkinetic, normal, decreased, absent)
Identification of suspected stricture | At the post-water ingestion scan 20-30 minutes after ingestion
  Identification of suspected stricture with documentation of changes post WICUS (measured luminal distension in millimeters)
Measurement of bowel wall thickness | At the post-water ingestion scan 20-30 minutes after ingestion
  Bowel wall thickness of the terminal ileum and any diseased segment (in millimeters)
Measurement of hyperaemia of the bowel wall of any diseased terminal ileal segment | At the post-water ingestion scan 20-30 minutes after ingestion
  Assessment of the bowel wall with colour doppler, and grading hyperaemia with the modified Limberg score (0 = no vascularity, 1 = localised vascularity, 2 = extensive vascularity, 3 = hyperemia extending into mesentery)
Pre-stenotic dilatation | At the post-water ingestion scan 20-30 minutes after ingestion
  Measurement of prestenotic luminal distension (in millimeters) proximal to any diseased terminal ileum segment
Diet effeect on the study | At the post-water ingestion scan 20-30 minutes after ingestion
  To determine if fasted patients (>2 hours no fluid and >3 hours no solid food [meal/snack/nothing]) were more likely to be included in the study due to lesser luminal distention
Global assessment as assessed by blinded assessors | At the post-water ingestion scan 20-30 minutes after ingestion
  Likert scale (5 point) global assessment 1-5 (1=Poor/inadequate views, 5=excellent view)
Distension assessment | At the post-water ingestion scan 20-30 minutes after ingestion
  Binary assessment of distension - either poor or adequate
Grade of peristalsis | At the post-water ingestion scan 20-30 minutes after ingestion
  Grade of peristalsis hyperkinetic / normal / decreased / absent

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Health, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No